CLINICAL TRIAL: NCT06087991
Title: Buprenorphine Induction and Naloxone Distribution Program-Combined With Warm Hand-Off Referral to Continued Treatment
Acronym: BINDeR-TX
Status: Completed | Type: Observational
Sponsor: Jerry Cochran (Other)
Responsible Party: Sponsor-Investigator, Jerry Cochran, Associate Professor, University of Utah
Organization: University of Utah (Other)
Other Study IDs: 158724
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Quantitative Interviews: Any Castleview patient who participates in this model will be emailed both the Patient Satisfaction Questionnaire Short Form (PSQ 18) and the Government Performance and Results Act surveys after hospital discharge, six months, and at discharge for buprenorphine.
  Interventions: Behavioral: Implementation of the BINDeR-Tx service model
- Qualitative Interviews: Qualitative interviews among providers, stakeholders and community members associated with Castleview Hospital will be conducted after the model has been deployed. The qualitative interviews will come from The Consolidated Framework for Implementation Research (CFIR) which is a validated tool that was developed that was developed to evaluate implementation studies.
  Interventions: Behavioral: Implementation of the BINDeR-Tx service model

INTERVENTIONS:
Behavioral: Implementation of the BINDeR-Tx service model — ED-initiated buprenorphine, discharge with naloxone, and warm-hand off referral for continued treatment for individuals with OUD. This is considered standard treatment at the University of Utah ED. In order to extend these services to rural hospitals this study will be assisting Castleview Hospital to establish a similar program.

SUMMARY:
This study is a collaboration between the University of Utah and Castleview Hospital in Price, Utah.

Buprenorphine is a medication approved by the FDA to treat Opioid Use Disorder (OUD). Castleview Hospital currently does not prescribe buprenorphine in the emergency department (ED) instead it refers patients to outside addiction treatment facilities. This is a service focused project which the University of Utah will provide mentoring and education to Castleview in implementing an in ED buprenorphine/naloxone distribution program along with referral to continued services. After the program has been implemented, the investigators will evaluate it using quantitative surveys of program participants and qualitative interviews of hospital staff and stakeholders.

DETAILED DESCRIPTION:
Among health care environments, ED often are the front lines of care for those with OUD or who experience opioid overdose.

The University of Utah Hospital ED has the Bridge Program which provides buprenorphine and naloxone with warm-hand off referral for continued treatment to people presenting with OUD. In order to extend the services offered by the Bridge Program to rural hospitals, the investigators will be providing mentoring and education to Castleview Hospital in establishing a similar program. Castleview Hospital is the only acute care hospital that serves Carbon and Emery counties, which outside of the Salt Lake City metro area have the highest opioid overdose rates in the State of Utah.

This project will utilize both quantitative and qualitative measures to evaluate the impact of this program on patients, hospital staff, and community members.

ELIGIBILITY:
Inclusion Criteria:

For qualitative interviews with providers, administrators, stakeholders:

* Must be affiliated with Castleview Hospital as a provider, administrator or stakeholder.

For the quantitative surveys:

* Must be a Castleview Hospital patient who receives the BINDeR-Tx model.

Exclusion Criteria:

For qualitative interviews with providers, administrators, stakeholders:

* Not familiar with the BINDeR-Tx model
* No interaction with the BINDeR-Tx model

For the quantitative surveys:

* Unable to speak and read English
* Subject is unable to provide contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 qualitative interviews of Castleview providers and stakeholders; 337 Castleview patient participants given buprenorphine and naloxone kits
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Patient Focused: Number of patients receiving services. | 24 months
  Will be the aggregate number of individuals who received ED-initiated buprenorphine.

SECONDARY OUTCOMES:
Implementation and service quality: Satisfaction with projected service | 24 months.
  Qualitative interviews including clinicians, hospital staff, and community members associated with Castleview Hospital will be the investigators using the Consolidated Framework for Implementation Research (CFIR).
Implementation and service quality: Patient satisfaction | enrollment and 6 months post enrollment
  Patient satisfaction will be assessed using the Patient Satisfaction Questionnaire Short Form (PSQ-18)
Substance use diagnosis and treatment | enrollment and 6 months post enrollment
  Using the Government Performance and Results Act (GPRA) Outcome questions on substance use within the past 30 days, other substance use disorder diagnoses and treatment in the past 30 days, and mental health diagnoses.
Social Connectedness | enrollment and 6 months post enrollment
  Social connectedness will be measured using the GPRA questions on mutual support group attendance in the last 30 days and relationship satisfaction and support.
Living Conditions | enrollment and 6 months post enrollment
  Living conditions will be measured using the GPRA questions on residence within the past 30 days.
Mental and Physical Health Problems and Treatment/Recovery | enrollment and 6 months post enrollment
  Mental and physical health problems and treatment/recovery will be measured using the GPRA questions on mental health symptoms and medical care received in the past 30 days and insurance status.
Legal Status | enrollment and 6 months post enrollment
  Legal status will be measured using the GPRA questions on incarceration in the past 30 days, charges, trial, sentencing, parole, probation, and drug court status.
Discharge status | enrollment and 6 months post enrollment
  Discharge status will be measured using the GRPA questions on substance use diagnosis and treatment in the past 30 days.
Follow-up Status | enrollment and 6 months post enrollment
  Follow-up status will be measured using the GPRA questions on contact and follow-up status.
Education, Employment, and Income | enrollment and 6 months post enrollment
  Education, employment, and income will be measured using the GPRA questions on education level, employment status, living expenses and income status.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cochran, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Seliski N, Madsen T, Eley S, Colosimo J, Engar T, Gordon A, Barnett C, Humiston G, Morsillo T, Stolebarger L, Smid MC, Cochran G. Implementation of a rural emergency department-initiated buprenorphine program in the mountain west: a study protocol. Addict Sci Clin Pract. 2024 Sep 3;19(1):63. doi: 10.1186/s13722-024-00496-0. PMID 39228007